CLINICAL TRIAL: NCT01758432
Title: A Randomized, Double-Blind, Vehicle-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered PRT064445 After Dosing to Steady State With One of Four Direct/Indirect fXa Inhibitors in Healthy Volunteers
Brief Title: Phase 2 Healthy Volunteer Study to Evaluate the Ability of PRT064445 to Reverse the Effects of Several Blood Thinner Drugs on Laboratory Tests (Module 1 of 4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-502 Module 1
Record Dates: First submitted 2012-12-18; First posted 2013-01-01 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — PRT064445; apixaban

STUDY DESIGN:
Intervention Model Description: This study has four modules with a total of 21 cohorts, each module was reported and submitted separately.
  Module 1, NCT01758432 (54 subjects with 7cohorts including placebo); Module 2, NCT03578146 (48 subjects with 6 cohorts including placebo); Module 3, NCT03551730 (27 subjects with 4 cohorts including placebo); Module 4, NCT03551743 (28 subjects with 4 cohorts including placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Module 1 (90 mg bolus) (Experimental): 90 mg PRT064445 given as a single IV
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 (210 mg bolus) (Experimental): 210 mg PRT064445 given as a single IV bolus
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 (420 mg bolus) (Experimental): 420 mg PRT064445 given as a single IV bolus
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 (420 mg bolus + 180 mg infusion) 4 mg/min (Experimental): 600 mg PRT064445 given as follows: 420 mg IV over ~14 minutes (~30 mg/min), followed by a continuous infusion of 180 mg (4 mg/min over 45 minutes)
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 (420 mg bolus + 180 mg bolus) 30mg/min (Experimental): 600 mg PRT064445 given as follows: up to 420 mg IV over ~14 minutes (~30 mg/min), followed by a second bolus of 180 mg IV over ~6 minutes (~30 mg/min), 45 minutes after completion of the bolus
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 (420 mg bolus + 480 mg infusion) 4mg/min (Experimental): 900 mg PRT064445 given as follows: 420 mg IV, followed by a continuous infusion of 480 mg (4 mg/min over 120 minutes
  Interventions: Combination Product: PRT064445/Apixaban; Combination Product: Placebo/Apixaban
- Module 1 Placebo (Placebo Comparator): Placebo administered intravenously (IV) as a bolus, two bolus doses or a bolus followed by continuous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: PRT064445/Apixaban
  Other Names: Andexanet
  Arms: Module 1 (210 mg bolus); Module 1 (420 mg bolus + 180 mg bolus) 30mg/min; Module 1 (420 mg bolus + 180 mg infusion) 4 mg/min; Module 1 (420 mg bolus + 480 mg infusion) 4mg/min; Module 1 (420 mg bolus); Module 1 (90 mg bolus)
Combination Product: Placebo/Apixaban
  Arms: Module 1 (210 mg bolus); Module 1 (420 mg bolus + 180 mg bolus) 30mg/min; Module 1 (420 mg bolus + 180 mg infusion) 4 mg/min; Module 1 (420 mg bolus + 480 mg infusion) 4mg/min; Module 1 (420 mg bolus); Module 1 (90 mg bolus)
Drug: Placebo
  Arms: Module 1 Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of PRT064445 to reverse the effects of several blood thinner drugs on laboratory tests. The study also is evaluating the blood levels of PRT064445 given at different doses.

DETAILED DESCRIPTION:
A randomized, double-blind, vehicle-controlled study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of intravenously administered PRT064445 after dosing to steady state with one of four direct/indirect fXa inhibitors in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 45 years old

Exclusion Criteria:

* History (including family history) or symptoms of, or risk factors for bleeding
* History (including family history) of or risk factors for a hypercoagulable or thrombotic condition
* Absolute/relative contraindication to anticoagulation or treatment with specific anticoagulants
* History of major surgery, severe trauma or bone fracture within 3 months prior to dosing; or planned surgery within 1 month after dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tempe, Arizona, United States

REFERENCES:
- [Derived] Siegal D, Lu G, Leeds JM, Karbarz M, Castillo J, Mathur V, Hutchaleelaha A, Sinha U, Kitt M, McClure M, Hollenbach SJ, Curnutte JT, Conley PB, Crowther M. Safety, pharmacokinetics, and reversal of apixaban anticoagulation with andexanet alfa. Blood Adv. 2017 Sep 22;1(21):1827-1838. doi: 10.1182/bloodadvances.2017007112. eCollection 2017 Sep 26. PMID 29296829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred at investigative site in the US between November 2012 through October 2013
Pre-assignment Details: Apixaban was administered orally at 5 mg twice daily for 6 days to steady-state in an open label fashion. Subjects were then randomized to receive study treatment (andexanet:placebo, 6:3) intravenously at different doses/dose regimens on Day 6, all bolus doses administered such that they ended at 3 hours after the last dose of apixaban.
Groups:
- Module 1 Placebo: Placebo was administered intravenously (IV) as a bolus, two bolus doses or a bolus followed by continuous infusion.
- Module 1 ( 90 mg): 90 mg andexanet IV bolus administered over 3 minutes (~30 mg/min)
- Module 1 (210 mg): 210 mg andexanet IV bolus administered over 10 minutes (~30 mg/min)
- Module 1 (420 mg): 420 mg andexanet IV bolus administered over 15 minutes (~30 mg/min)
- Module 1 (420 mg Bolus + 180 mg Infusion): 420 mg andexanet IV bolus administered over ~14 minutes (~30 mg/min) followed immediately by a 180 mg continuous IV infusion (4 mg/min over 45 minutes) [total 600 mg]
- Module 1 (420 mg Bolus + 180 mg Bolus): 420 mg andexanet/placebo IV bolus administered over ~14 minutes (~30 mg/min) followed after 45 minutes by a second bolus of 180 mg over~ 6 minutes (~30 mg/min) [total 600 mg]
- Module 1 (420 mg Bolus + 480 mg Infusion): 420 mg andexanet IV bolus administered over ~14 minutes (~30 mg/min) followed immediately by a 480 mg continuous IV infusion (4 mg/min over 2 hours) [total 900 mg]
Period: Overall Study
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Started | 18 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 18 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 54 subjects were enrolled in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion) | Total
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] — 54 subjects were enrolled in this study.
  years | 33.4 (7.69) | 33.7 (8.48) | 35.0 (7.32) | 33.8 (5.78) | 31.7 (9.50) | 32.5 (8.60) | 31.8 (6.97) | 33.2 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 8
  Male | 17 | 6 | 5 | 6 | 3 | 3 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent Change From Baseline in Anti-fXa Activity at 2 Mins Following Andexanet/Placebo Administration
Description: Anti-fXa activity was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Anti-fXa activity was measured using a commercial kit (Coamatic Heparin-82 33 9363, DiaPharma)
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 54 subjects who received andexanet or placebo were included in the pharmacodynamics (PD) analysis
Measure: Mean (Standard Deviation); unit: Percent change in anti-fXa activity
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
Percent change in anti-fXa activity | -7.06 (10.801) | -67.79 (7.731) | -78.51 (3.815) | -95.04 (1.375) | -94.03 (1.870) | -93.07 (1.765) | -92.82 (1.267)
Statistical Analysis 1: Comparison: Module 1 Placebo vs Module 1 ( 90 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -95.74
Statistical Analysis 2: Comparison: Module 1 Placebo vs Module 1 (210 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -130.5
Statistical Analysis 3: Comparison: Module 1 Placebo vs Module 1 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -129.86
Statistical Analysis 4: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -165.91
Statistical Analysis 5: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Bolus); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -167.94
Statistical Analysis 6: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 480 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -135.91

2. Secondary Outcome: Efficacy: Percent Change From Baseline in Thrombin Generation at 2 Mins Following Andexanet/Placebo Administration
Description: Thrombin generation was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Thrombin generation was measured using a TF-initiated thrombin generation assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 45 subjects who received andexanet or placebo were included in the PD analysis
Measure: Mean (Standard Deviation); unit: Percent change in thrombin generation
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
Percent change in thrombin generation | 28.11 (36.871) | 76.58 (47.729) | 137.50 (67.528) | 120.95 (91.301) | 222.56 (95.671) | 196.29 (65.406) | 191.77 (122.385)
Statistical Analysis 1: Comparison: Module 1 Placebo vs Module 1 ( 90 mg); Test type: Superiority; p = 0.0004, ANCOVA; Least Squares Means (Difference) = 85559.49
Statistical Analysis 2: Comparison: Module 1 Placebo vs Module 1 (210 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 105508.3
Statistical Analysis 3: Comparison: Module 1 Placebo vs Module 1 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 182753.2
Statistical Analysis 4: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 193684.5
Statistical Analysis 5: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Bolus); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 178055
Statistical Analysis 6: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 480 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = 169709.9

3. Secondary Outcome: Efficacy: Percent Change From Baseline in Unbound Apixaban Plasma Concentration at 2 Mins Following Andexanet/Placebo Administration
Description: Unbound apixaban concentrations was measured immediately prior to (Baseline) and at 2 mins following andexanet/placebo administration. Unbound plasma concentrations for apixaban were determined by a rapid equilibrium dialysis method followed by Liquid Chromatography-Mass Spectometry assay.
Time Frame: Baseline to 2 minutes following the end of andexanet/placebo administration
Population: 54 subjects who received apixaban were included in the apixaban pharmacokinetics (PK) analysis
Measure: Mean (Standard Deviation); unit: % change in unbound apixaban concentrat.
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
% change in unbound apixaban concentrat. | -5 (14) | -51 (12) | -54 (7) | -72 (7) | -79 (6) | -89 (3) | -84 (6)
Statistical Analysis 1: Comparison: Module 1 Placebo vs Module 1 ( 90 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -4.58
Statistical Analysis 2: Comparison: Module 1 Placebo vs Module 1 (210 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -4.29
Statistical Analysis 3: Comparison: Module 1 Placebo vs Module 1 (420 mg); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -6.15
Statistical Analysis 4: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -6.79
Statistical Analysis 5: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 180 mg Bolus); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -7.49
Statistical Analysis 6: Comparison: Module 1 Placebo vs Module 1 (420 mg Bolus + 480 mg Infusion); Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Means (Difference) = -6.71

4. Secondary Outcome: Andexanet Maximum Observed Plasma Concentration (Cmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Cmax was taken directly from the raw data.
Time Frame: Blood was collected at predose, 0.033, 0.2, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6.5, 7.5, 8.5 and 14.5 hours postdose.
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | NA (NA) — Andexanet not administered (placebo group) | 21200 (2400) | 42800 (5620) | 81400 (10900) | 93300 (18400) | 88000 (9010) | 90800 (29600)

5. Secondary Outcome: Andexanet Time of Maximum Observed Plasma Concentration (Tmax)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Tmax was taken directly from the raw data.
Time Frame: as for outcome 4
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Median (Full Range); unit: hr
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
hr | NA [NA to NA] — Andexanet was not administered (placebo group) | 0.07 [0.07 to 0.08] | 0.15 [0.14 to 0.30] | 0.27 [0.26 to 0.29] | 0.43 [0.25 to 0.52] | 0.27 [0.26 to 0.31] | 0.28 [0.272 to 0.29]

6. Secondary Outcome: Andexanet Total Volume of Distribution (Vss)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. Vss was calculated using a non-compartmental approach.
Time Frame: as for outcome 4
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
L | NA (NA) — Andexanet not administered (placebo group) | 6.97 (1.42) | 6.18 (1.31) | 6.26 (0.742) | 5.11 (1.64) | NA (NA) — Vss calculations do not take into account the 45 minute intervals between doses. | 4.01 (0.951)

7. Secondary Outcome: Andexanet Area Under the Drug Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf )
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. AUC0-inf was calculated using a non-compartmental approach
Time Frame: as for outcome 4
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | NA (NA) — Andexanet was not administered (placebo group) | 23400 (3460) | 49200 (3960) | 93500 (15500) | 131000 (20500) | 155000 (16200) | 213000 (33900)

8. Secondary Outcome: Andexanet Total Systemic Clearance (CL)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electrochemiluminescent assay. CL was calculated using a non-compartmental approach, calculated as Dose/AUC0-inf
Time Frame: as for outcome 4
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
L | NA (NA) — Andexanet not administered (placebo group) | 3.93 (0.634) | 4.29 (0.331) | 4.60 (0.814) | 4.70 (0.887) | NA (NA) — Not determined as CL | 4.30 (0.608)

9. Secondary Outcome: Andexanet Apparent Terminal Elimination Half-life (t1/2)
Description: Plasma concentrations of andexanet was determined using a validated method that involved analysis of citrated human plasma by an electro chemiluminescent assay. t1/2 was determined by linear regression of the log concentration on the terminal portion of the plasma concentration-time curve.
Time Frame: as for outcome 4
Population: 36 subjects who received andexanet were included in the andexanet PK analysis
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Number analyzed (Participants) | 18 | 6 | 6 | 6 | 6 | 6 | 6
hr | NA (NA) — Andexanet was not administered (placebo group) | 5.51 (0.84) | 5.12 (1.66) | 5.02 (2.02) | 4.35 (1.40) | 5.79 (2.00) | 6.45 (0.41)

ADVERSE EVENTS:
Time Frame: ~7 weeks
Description: Only subjects who received at least one dose of study drug were included in the safety analysis.
Groups:
- Module 1 (210 mg): 210 mg andexanet IV bolus administered over 10 minutes (~30 mg/min) 420 mg andexanet IV bolus administered over 15 minutes (~30 mg/min)
Arm/Group | Module 1 Placebo | Module 1 ( 90 mg) | Module 1 (210 mg) | Module 1 (420 mg) | Module 1 (420 mg Bolus + 180 mg Infusion) | Module 1 (420 mg Bolus + 180 mg Bolus) | Module 1 (420 mg Bolus + 480 mg Infusion)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 14/18 | 3/6 | 3/6 | 5/6 | 4/6 | 2/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Module 1 Placebo (N=18) | Module 1 ( 90 mg) (N=6) | Module 1 (210 mg) (N=6) | Module 1 (420 mg) (N=6) | Module 1 (420 mg Bolus + 180 mg Infusion) (N=6) | Module 1 (420 mg Bolus + 180 mg Bolus) (N=6) | Module 1 (420 mg Bolus + 480 mg Infusion) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemmia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site pain (General disorders) | 4 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site paraesthesia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 1 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Conducted in healthy volunteers at Clinical Research Organization